CLINICAL TRIAL: NCT06717802
Title: Endometrial Receptivity Prediction During in Vitro Fertilization Using Artificial Intelligence Analysis of Vaginal Ultrasound Images
Brief Title: Endometrial Receptivity Prediction During in Vitro Fertilization Using Artificial Intelligence
Status: Recruiting | Type: Observational
Sponsor: Gottsegen National Cardiovascular Institute (Other)
Collaborators: Dunamenti REK Reprodukcios Kozpont (Unknown)
Responsible Party: Principal Investigator, Márton Kolossváry, Head of Education and Research, Gottsegen National Cardiovascular Institute
Other Study IDs: endoAI
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Infertility; Infertility (IVF Patients)
Keywords: assisted reproduction; Artificial intelligence (AI); Endometrial receptivity; Embryo implantation; Ultrasound imaging
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to use artificial intelligence to analyse vaginal ultrasound images of the uterine lining (endometrium) taken during routine IVF treatment, which may predict implantation success during IVF treatment.

Participation in the study is voluntary, involves no additional testing or intervention beyond routine procedures, and consent can be withdrawn verbally or in writing at any time without cause or adverse consequences.

Over a three-year period, the trial is expected to enrol approximately 1,500 patients between the ages of 18 and 40 who are indicated for IVF treatment and who volunteer for treatment.

Patients enrolled in the study will not be required to attend more clinic visits during treatment than they would otherwise have to. During the trial, certain patient-specific data (age, indication for treatment, body mass index), stimulation-specific data (duration of stimulation, type and dose of drug, endometrial thickness), ultrasound scans and outcome-specific data (treatment failure, biochemical pregnancy, clinical pregnancy) will be collected. The data will be stored in a secure database. The data collected during the study will only be accessible to the professionals involved in the study and no information, including personal data, will be disclosed to third parties.

DETAILED DESCRIPTION:
Infertility affects one in six people globally over the duration of their reproductive lives. For successful IVF treatment, three essential things are needed: a euploid embryo, receptive endometrium and in case of frozen embryos, the exact timing of the transfer. Several methods are available for evaluating embryos, such as: microscopic evaluation (e.g. Gardner grade), genetic tests (PGT), biochemical tests (non-invasive PGT). Furthermore, morphological and morphokinetic evaluation is possible using time-lapse video surveillance systems that are evaluated using artificial intelligence. The most common method for testing the receptivity of the endometrium is the determination of the largest diameter measured in the mid-sagittal plane. A thickness between 7 and 10 mm is considered the cut-off for successful implantation. Further studies were conducted on the level of the serum and endometrial progesterone, the volume, echogenicity, peristalsis of the endometrium, the flow conditions in it and the success of implantation. The predictive value of hysteroscopy, 3D ultrasound and the role of ultrasound elastography to predict pregnancy outcome has been investigated. The above-mentioned tests for endometrial receptivity have not been widely used in practice, and there is currently no method for predicting endometrial receptivity in everyday practice.

As the quality of imaging has improved, the focus has shifted to analyzing the pattern of the endometrium, the latest research using artificial intelligence.

The aim of this study is to investigate whether segmentation and analysis of the endometrium using artificial intelligence in vaginal ultrasound images taken during stimulation and on the day of transfer can help to more accurately determine the receptivity of the endometrium. The significance of this is that in case of poor implantation chances it is possible to freeze the embryo(s) and have the opportunity to implant the embryo in a subsequent natural or hormone replacement therapy cycle, possibly with better chances.

ELIGIBILITY:
Inclusion Criteria:

* Female patient 18-40 years, for whom IVF is indicated
* Maximum 3 unsuccessful previous embryo transfers
* Only cycles in which single blastocyst is transferred

Exclusion Criteria:

* Congenital uterine anomalies, fibroids, adenomyosis, Asherman-syndrome or any other conditions resulting in malformation of the uterus
* Presence of hydrosalpinx
* Endometriosis
* Planned freeze-all cycle
* Positive hepatitis B, hepatitis C or HIV screening test

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who volunteer for IVF treatment at participating infertility centres
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy | The date of the ultrasound confirmed clinical pregnancy scheduled at 28 days following embryo transfer
  Clinical pregnancy: pregnancy can be confirmed through ultrasound visualization of the gestational sac or heartbeat

CONTACTS AND LOCATIONS:
Locations (1):
- Dunamenti REK Reprodukcios Kozpont, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided